CLINICAL TRIAL: NCT06188351
Title: A Prospective, Multicenter, Randomized, Controlled Trial to Evaluate the Safety and Efficacy of a Three Dimensional Navigation Intracardiac Guidance Kit for Atrial Septal Puncture
Brief Title: Three Dimensional Navigation IntraCardiac Guidance Kit for Atrial Septal Puncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Wuhan Greenrhythm Medical Technology Co., LTD (Industry)
Responsible Party: Principal Investigator, Yan Wang, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3DASP study
Record Dates: First submitted 2023-11-19; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial septal puncture; Three dimensional; fluroscopy; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three-Dimensional Navigation Atrial Septal Puncture (Experimental): Atrial septal puncture will be performed using a three-dimensional navigation intracardiac guidance kit
  Interventions: Device: Three-Dimensional Navigation Atrial Septal Puncture
- Conventional Atrial Septal Puncture (Active Comparator): Atrial septal puncture will be performed using trational atrial septal puncture kit using traditional method.
  Interventions: Device: Conventional Atrial Septal Puncture

INTERVENTIONS:
Device: Three-Dimensional Navigation Atrial Septal Puncture — Atrial septal puncture will be performed using a three-dimensional navigation intracardiac guidance kit
  Arms: Three-Dimensional Navigation Atrial Septal Puncture
Device: Conventional Atrial Septal Puncture — Atrial septal puncture will be performed using traditioanl two-dimensional atrial septal puncture kit using traditional method.
  Arms: Conventional Atrial Septal Puncture

SUMMARY:
This study aims to evaluate the safety and efficacy of a three-dimensional navigation intracardiac guidance kit to perform atrial septal puncture in patients requiring catheter ablation, which will be compared with procedures using traditional kit for atrial septal puncture.

DETAILED DESCRIPTION:
Atrial septal puncture has become a key technique in cardiac interventional procedures. Traditional septal punctures are routinely perfomed under two-dimensioanl guidance, whic are likely to be not acurate sometimes.

This study is aimed to study the safety and efficacy of a novel designed three-dimensional navigation Intracardiac guidance kit for atrial septal puncture in patients with atrial fibrillation requiring catheter ablation and to explore the possibility of transseptal without fluoroscopy using the three-dimensional positioning intracardiac guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with atrial fibrillation.
2. Requiring catheter ablation therapy.
3. Voluntarily sign the informed consent.

Exclusion Criteria:

1. Previous atrial septal puncture.
2. Blood clots in the left atrium or left atrial appendage
3. Left atrial mucinous tumor.
4. Atrial septal defect, including previous surgical correction or interventional occlusion.
5. Acute or severe systemic infection.
6. Cardiac function (NYHA classification) Ⅲ-Ⅳ.
7. Contraindications to anticoagulation.
8. Left ventricular ejection fraction <35%.
9. Patients with untreated or uncontrolled hyperthyroidism or hypothyroidism.
10. Patients with malignancy with expected survival of less than 1 year.
11. Myocardial infarction or any cardiac intervention or open procedure within the last 3 months
12. Stroke and other cerebrovascular disease or thromboembolic disease within the last 3 months.
13. Participated in clinical trials of other drugs or devices in the past 3 months.
14. Any other condition that the investigator deems inappropriate for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of atrial septal puncture | one day
  Successful atrial septal puncture is defined as the right and left interatrial pathways are established and the ablation catheter can enter the left atrium smoothly for subsequent ablation operations.
X-Ray exposure time | one day
  X-ray exposure time from the successful femoral vein puncture to the entry of the external sheath into the left atrium (ending with heparin saline flushing of the sheath).

SECONDARY OUTCOMES:
First puncture success rate of atrial septum | one day
  When the first septal puncture is performed, the puncture sheath is passed through the septal puncture from the right atrium into the left atrium.
Atrial septal puncture duration | one day
  Time taken from the time the puncture needle enters the dilator to the time when heparin saline is applied to flush the sheath after the external sheath enters the left atrium.
Total operation time | one day
  Time taken from the start of successful femoral vein puncture to the entry of the external sheath into the left atrium (ending with heparin saline flushing of the sheath).
Performance evaluation of a three-dimensional positioning intracardiac guidance kit | one day
  The investigators evaluated the products in terms of pushing performance, retraction performance, torsional control performance, bending resistance/kinking resistance in dilator, catheter sheath, and blood; and tracking performance of the guidewire, catheter sheath, and puncture needle in the 3D calibration system, respectively.

OTHER OUTCOMES:
（Incidence (%) and frequency (number of events) of (serious) adverse events | one day
  （Incidence (%) and frequency (number of events) of (serious) adverse events.
Incidence (%) and frequency (number of events) of device-related (serious) adverse events | one day
  Incidence (%) and frequency (number of events) of device-related (serious) adverse events.
Incidence of device defects and number of events that occurred | one day
  Incidence of device defects and number of events that occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, PhD, Principal Investigator — Tongji Hospital Wuhan, Hubei China
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu R, Liu N, Lu J, Zhao X, Hu Y, Zhang J, Xu F, Tang R, Bai R, Akar JG, Dong J, Ma C. 3-Dimensional Transseptal Puncture Based on Electrographic Characteristics of Fossa Ovalis: A Fluoroscopy-Free and Echocardiography-Free Method. JACC Cardiovasc Interv. 2020 May 25;13(10):1223-1232. doi: 10.1016/j.jcin.2020.03.015. PMID 32438994
- [Background] Graham AJ, Honarbakhsh S, O'Brien B, Schilling RJ. A Simplified Trans-Septal Puncture Technique using a Needle Free Approach for Cryoablation of Atrial Fibrillation. J Atr Fibrillation. 2017 Aug 31;10(2):1628. doi: 10.4022/jafib.1628. eCollection 2017 Aug-Sep. PMID 29250235
- [Background] Hang F, Cheng L, Liang Z, Dong R, Wang X, Wang Z, Wang Z, Wu Y. Study on the Curative Effect and Safety of Radiofrequency Catheter Ablation of Paroxysmal Atrial Fibrillation via Zero-Fluoroscopy Transseptal Puncture under the Dual Guidance of Electroanatomical Mapping and Intracardiac Echocardiography. Cardiol Res Pract. 2021 May 24;2021:5561574. doi: 10.1155/2021/5561574. eCollection 2021. PMID 34123417
- [Background] Fromentin S, Sarrazin JF, Champagne J, Nault I, Philippon F, Molin F, Blier L, O'Hara G. Prospective comparison between conventional transseptal puncture and transseptal needle puncture with radiofrequency energy. J Interv Card Electrophysiol. 2011 Sep;31(3):237-42. doi: 10.1007/s10840-011-9564-2. Epub 2011 Apr 19. PMID 21503731
- [Background] Knecht S, Jais P, Nault I, Wright M, Matsuo S, Madaffari A, Lellouche N, O'Neill MD, Derval N, Deplagne A, Bordachar P, Sacher F, Hocini M, Clementy J, Haissaguerre M. Radiofrequency puncture of the fossa ovalis for resistant transseptal access. Circ Arrhythm Electrophysiol. 2008 Aug;1(3):169-74. doi: 10.1161/CIRCEP.108.788000. Epub 2008 Jun 23. PMID 19808411
- [Background] Sawhney V, Breitenstein A, Watts T, Garcia J, Finlay M, Lowe M, Hunter R, Earley MJ, Schilling RJ, Sporton S, Dhinoja M. A novel technique for performing transseptal puncture guided by a non-fluoroscopic 3D mapping system. Pacing Clin Electrophysiol. 2019 Jan;42(1):4-12. doi: 10.1111/pace.13541. Epub 2018 Nov 28. PMID 30397922
- [Background] Koektuerk B, Yorgun H, Koektuerk O, Turan CH, Gorr E, Horlitz M, Turan RG. Rotational Angiography Based Three-Dimensional Left Atrial Reconstruction: A New Approach for Transseptal Puncture. Cardiovasc Ther. 2016 Feb;34(1):49-56. doi: 10.1111/1755-5922.12167. PMID 26607305
- [Background] Manolis AS. Transseptal Access to the Left Atrium: Tips and Tricks to Keep it Safe Derived from Single Operator Experience and Review of the Literature. Curr Cardiol Rev. 2017;13(4):305-318. doi: 10.2174/1573403X13666170927122036. PMID 28969539
- [Background] Rodriguez-Manero M, Martinez-Sande JL, Fandino R, Garcia-Seara J, Chierchia GB, Fernandez-Lopez XA, Osorio I, de Alegria AM, Souto-Bayarri M, Brugada P, Gonzalez-Juanatey JR. Fluoroscopic integration of the cardiac computed tomography as a guide for transseptal puncture during atrial fibrillation ablation: A feasibility study. Int J Cardiol. 2015 Apr 1;184:274-275. doi: 10.1016/j.ijcard.2015.02.035. Epub 2015 Feb 24. No abstract available. PMID 25731834
- [Background] Li C, Zhang J, Li S, Sang C, Liu N, Du X, Dong J, Ma C. A novel and easy approach to difficult transseptal puncture during atrial fibrillation ablation. J Interv Card Electrophysiol. 2021 Nov;62(2):269-276. doi: 10.1007/s10840-020-00891-y. Epub 2020 Oct 9. PMID 33034794
- [Background] ROSS J Jr, BRAUNWALD E, MORROW AG. Transseptal left atrial puncture; new technique for the measurement of left atrial pressure in man. Am J Cardiol. 1959 May;3(5):653-5. doi: 10.1016/0002-9149(59)90347-9. No abstract available. PMID 13649591
- [Background] Vlastra W, Delewi R, Sjauw KD, Beijk MA, Claessen BE, Streekstra GJ, Bekker RJ, van Hattum JC, Wykrzykowska JJ, Vis MM, Koch KT, de Winter RJ, Piek JJ, Henriques JPS. Efficacy of the RADPAD Protection Drape in Reducing Operators' Radiation Exposure in the Catheterization Laboratory: A Sham-Controlled Randomized Trial. Circ Cardiovasc Interv. 2017 Nov;10(11):e006058. doi: 10.1161/CIRCINTERVENTIONS.117.006058. PMID 29089313
- [Background] Salghetti F, Sieira J, Chierchia GB, Curnis A, de Asmundis C. Recognizing and reacting to complications of trans-septal puncture. Expert Rev Cardiovasc Ther. 2017 Dec;15(12):905-912. doi: 10.1080/14779072.2017.1408411. Epub 2017 Nov 30. PMID 29161923